CLINICAL TRIAL: NCT07167485
Title: Sleep Quality of Intensive Care Patients During Their Care Pathway.
Brief Title: Sleep Quality of Intensive Care Patients
Acronym: Réa-SLEEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/294/OB; 2020-A02632-37 (Other: ANSM)
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-05

CONDITIONS: Sleep Quality in Adult ICU Patients
Keywords: Detoxification and rehabilitation unit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of sleep quality — Sleep quality will be assessed each night in intensive care using a Richards-Campbell sleep questionnaire and an intensive care sleep questionnaire, completed by the patient.

SUMMARY:
Sleep deprivation is common in intensive care. Impaired sleep quality and quantity and altered circadian rhythms have been observed. Polysomnography is the gold standard for sleep analysis. However, it is difficult to perform due to technical constraints and the lack of a consensus definition of the different stages of sleep for intensive care patients. Alternative methods to polysomnography would be useful for better defining sleep disturbances. There are many factors that can disrupt sleep, including environmental disturbances, sedative drugs, mechanical ventilation, and the severity of the condition that led to the patient's admission to intensive care. The consequences of this deprivation include immune system disorders, neuropsychiatric disorders, and impaired functional recovery. Therapeutic management is currently limited, as no drug treatments have been shown to improve sleep quality. Furthermore, no ventilation method has been proven effective in improving sleep. Finally, regulating environmental disturbances-aiming to reduce light exposure, limit noise, and respect day/night rhythms-could improve sleep in intensive care patients. According to recent data, individual measures such as protective eye masks and earplugs have not improved patients' sleep architecture. The aim of our study is therefore to highlight the benefits of the withdrawal and rehabilitation unit (USR) in improving the quality of sleep in intensive care patients. The quality of sleep in intensive care patients in our department will be assessed using a questionnaire validated for intensive care patients, the Richard-Campbell questionnaire (RCSQ). We will also analyse various known risk factors for sleep disturbance in intensive care and USR patients.

DETAILED DESCRIPTION:
The research hypothesis is that the withdrawal and rehabilitation unit, thanks to its spatial organisation, admission policy, management of environmental disturbances and ventilation techniques, could be conducive to better sleep quality.

Patients with prolonged stays (≥14 days) account for between 4 and 11% of admissions to intensive care. By definition, intensive care is a place where patients may experience psychological distress and physical pain. Anxiety and depression, sleep disorders, disruption of the circadian rhythm and sleep debt frequently occur during a stay in intensive care and can hinder the patient's recovery. Measures that are simple in theory, aimed at promoting well-being, are sometimes very difficult to implement in such an acute care setting. Consequently, patients whose stay in intensive care is prolonged, whose clinical condition is stable but who still require 'intensive' care, particularly in relation to mechanical ventilation, muscle weakness and limited autonomy, will require control of these sources of psychological and physical suffering in the hope of promoting their well-being and even improving their rehabilitation. In intensive care, the main sources of discomfort are related to the environment (noise and excessive light) or work organisation, but also to more or less invasive care procedures: procedures associated with ventilation (tracheal suction, extubation), repeated blood sampling, catheter insertion, patient positioning in bed (pain associated with immobilisation, change of position, etc.). Numerous studies report very high noise levels in intensive care units, well above the recommended levels of 45 dB, due to alarms, equipment (ventilators, nebulisers, etc.), the behaviour of paramedical staff, and also medical staff (peaks during visits). An interesting alternative may then be to transfer the patient to a specific unit, either for weaning and rehabilitation or for continuous post-resuscitation care.

In Rouen, for example, there is a respiratory weaning and rehabilitation unit with specialised nursing staff in an environment considered more conducive to weaning and rehabilitation (specific paramedical team, daytime activities, no night-time admissions, corridor lights turned off at night, reasoned monitoring of vital signs). This unit could also be conducive to better control of environmental disturbances to ensure normal circadian rhythms and sufficient quantity and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* clinically stable (no amines or sedation for more than 48 hours)
* hospitalised for more than 7 days in intensive care
* conscious
* with no central neurological pathology
* with no major cognitive impairment
* with no sleep disorder (OSA, insomnia, restless legs syndrome)

Exclusion Criteria:

Age < 18 years old Patient refusal Person deprived of liberty by administrative or judicial decision or protected adult (under guardianship or trusteeship); Patient unable, for whatever reason, to read, understand or answer questionnaires (visual impairment, psychiatric or cognitive disorders, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care patients
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Assessing the quality of sleep in intensive care patients over time | At enrollment visit and Day 14
  Sleep quality according to the Richard-Campbell questionnaire (RCSQ) score. The Richards Campbell Sleep Questionnaire is a widely used sleep quality instrument comprising visual analogue scales (VAS) 0-100 mm allowing assessment of sleep depth, falling asleep, number of awakenings, percent of time awake, and overall quality of sleep domains. The higher the score, the better the quality of sleep.

SECONDARY OUTCOMES:
Compare sleep recovery rates according to hospital unit (intensive care or withdrawal and rehabilitation unit, USR). | At enrollment visit and Day 14
  The intensive care sleep questionnaire is a tool used to assess sleep quality. It includes visual analogue scales (VAS) from 0 to 100 mm that allow the depth of sleep, the time taken to fall asleep, the number of times the patient wakes up, the percentage of time spent awake and the overall quality of sleep to be assessed. It includes visual analogue scales (VAS) from 0 to 4 mm that assess difficulty falling asleep and difficulty staying asleep. The higher the score, the better the sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.